CLINICAL TRIAL: NCT03221192
Title: Qualitative Research to Characterize the Patient Experience of Nasal Polyps
Brief Title: Qualitative Analysis of Subject Experience of Nasal Polyps
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 206325
Record Dates: First submitted 2017-07-05; First posted 2017-07-18 (Actual); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Nasal Polyps
Keywords: Real-time data capture; Concept elicitation; Nasal polyps; Cognitive debriefing; Patient-reported outcomes; HRQoL
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects participating in CE and CD interviews: Twenty adult subjects from the US and 10 adult subjects from Germany with severe recurrent nasal polyps who have received nasal polyp surgery in the past 10 years prior to screening will be asked to participate in CE and CD interviews
  Interventions: Other: VAS questionnaire; Other: SNOT-22 questionnaire
- Subjects participating in interview and real-time data capture: Ten subjects from the US with severe recurrent nasal polyps who are participating in CE and CD interviews will be asked to complete the real-time data capture app task.
  Interventions: Other: VAS questionnaire; Other: SNOT-22 questionnaire; Other: Data capture app

INTERVENTIONS:
Other: VAS questionnaire — VAS questionnaire is a PRO tool in which subjects will be asked to evaluate overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 centimeter (cm) or 100 millimeter (mm) whereby 0 represents 'no symptom' and '10 or 100 represents 'as bad as you can imagine', Scores of 0-3 (or 0-30) are defined as mild disease, >3-7 (or >30-70) as moderate disease and >7-10 (or >70-100) as severe disease.
Other: SNOT-22 questionnaire — SNOT-22 is a PRO tool to measure HRQoL associated with rhinosinusitis with or without nasal polyps. It contains 22 nose, sinus, and general HRQoL items and subjects will be required to score the experience on a 6-point scale ranging from 0 (no problem) to 5 (Problem as bad as it can be) and identify the five most important items affecting their health.
Other: Data capture app — Real time data capture app is a smart-phone or web-based application which will allow the subjects to communicate about their experience of nasal polyps in real-time as they go about their daily lives via varying video, audio, photographic and text responses.
  Groups: Subjects participating in interview and real-time data capture

SUMMARY:
Nasal polyposis is a chronic inflammatory disease of the nose and sinuses. GlaxoSmithKline (GSK) is embarking on a clinical program to assess treatment of severe, recurrent nasal polyps with an anti-interleukin-5 (anti-IL5) (mepolizumab). Subject specific symptomatic endpoints will form the basis for the assessment of treatment benefit of nasal polyp therapies. However, there is a lack of published qualitative data regarding nasal polyps to understand the symptoms or health-related quality of life (HRQoL) impacts. This cross-sectional qualitative study aims to address this unmet gap by conducting semi-structured combined concept elicitation (CE) and cognitive debriefing (CD) telephone interviews and real-time data capture. The combined CE and CD interviews (each 90 minutes in duration) will investigate the subject experience of nasal polyps, and the relevance and understanding of existing patient-reported outcomes (PRO) instruments. The real-time data capture conducted over a 10 day period, will investigate the subject experience of the symptoms, HRQoL impacts and treatment of nasal polyps and any day-to-day variability that exists in these experiences in 'real time'. Twenty adult subjects in the United States (US), and 10 adult subjects in Germany with severe, recurrent nasal polyps will participate in the CE and CD interviews section of the study and of these, 10 subjects from US will also complete real-time data capture app task.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of bilateral nasal polyps as diagnosed by endoscopy or CT scan.
* Subject is aged 18 or over.
* Subject has severe nasal polyps symptoms defined as a subject-reported nasal obstruction VAS score of >5.
* Subject had at least one previous surgery in the past ten years for the removal of nasal polyps. Surgery in this case is defined as any procedure involving instruments with resulting incision and removal of polyp tissue from the nasal cavity (polypectomy).
* Subject is currently an eligible candidate for polypectomy defined by an overall subject-reported VAS symptom score of >7 and an endoscopic bilateral nasal polyp score of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity).
* Subject has symptoms consistent with chronic rhinosinusitis.
* Subject is currently receiving intranasal corticosteroids for the management of their nasal polyps.
* Subject is willing to participate in the study and provide informed consent.
* Subject is an English speaker and is able to read, write and fully understand the English language.
* Subject is willing to and able to attend and participate in a 90-minute interview to discuss their experiences of nasal polyps and obtain their feedback on several symptom/impact questionnaires.

For real-time data capture:

* Subject owns/or has access to either a smartphone [iPhone Operating System (iOS) or android] or tablet which has video, audio/microphone and photographic capabilities and access to either the Apple app store or Google play store to download the app.
* Subject is willing and able to take part in the real-time data application task and respond to a series of questions/tasks fielded to them via the application over the course of 10 days and is willing to respond to some brief questions following the real-time data capture task about their experience of using the app and completing the tasks, either during their interview or in a 5-10 minute telephone call following completion of the task.
* Subject would feel comfortable recording short videos of themselves and providing audio commentary in response to questions/tasks.

Exclusion Criteria:

* Subject has a diagnosis of cystic fibrosis.
* Subject has a diagnosis of eosinophilic granulomatosis with polyangiitis (also known as Churg Strauss syndrome), Young's, Kartagener's or dyskinetic ciliary syndromes).
* Subject has a diagnosis of antrochoanal polyps.
* Subject has a diagnosis of nasal septal deviation occluding one nostril.
* Subject has had acute sinusitis or upper respiratory tract infection in the last two week.
* Subject has ongoing rhinitis medicamentosa (rebound or chemical induced rhinitis).
* Subject has had an asthma exacerbation requiring admission to hospital in the last four weeks.
* Subject is currently or has previously taken part in a clinical trial for nasal polyps.
* Subject is unwilling or unable to comply with the requirements of the study or has a physical or mental condition or learning difficulties that, in the opinion of the physician, may affect the subject's ability to participate in the study, the responses he/she might provide or their ability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty adult subjects in the US, and 10 adult subjects in Germany with severe, recurrent nasal polyps who have undergone nasal polyp surgery in the past 10 years prior to screening will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gater A, Tolley C, Williams-Hall R, Trennery C, Bradley H, Sikirica MV, Nelsen L, Sousa AR, Bratton DJ, Chan R, von Maltzahn R. Patient-Reported Outcome Measures for Severe Recurrent Bilateral Nasal Polyps: Psychometric Evaluation and Content Validity. OTO Open. 2023 Dec 21;7(4):e84. doi: 10.1002/oto2.84. eCollection 2023 Oct-Dec. PMID 38130916
- [Derived] Hall R, Trennery C, Chan R, Gater A, Bradley H, Sikirica MV, von Maltzahn R, Sousa AR, Nelsen LM. Understanding the Patient Experience of Severe, Recurrent, Bilateral Nasal Polyps: A Qualitative Interview Study in the United States and Germany. Value Health. 2020 May;23(5):632-641. doi: 10.1016/j.jval.2019.11.005. Epub 2020 Mar 11. PMID 32389229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cross-sectional qualitative study to characterize the participants experience of nasal polyps. Participants were identified via partner recruitment agencies for participation in the Concept Elicitation (CE) or Cognitive Debriefing (CD) interview.
Pre-assignment Details: A total of 27 participants with severe, recurrent nasal polyps who underwent at least one nasal polyp surgery in the past 10 years were enrolled in the study. The study was conducted in the United States and Germany.
Groups:
- Interview Participants With Nasal Polyps: Participants with severe, recurrent nasal polyps who underwent at least one nasal polyp surgery in the past 10 years were enrolled.
Period: Overall Study
Arm/Group | Interview Participants With Nasal Polyps
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: Years] | 48.4 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  Black/African American | 2
  Hispanic | 4
  Asian/Pacific islander | 1
  Multiple | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Primary Symptoms
Description: During the CE section of the interview, participants were asked a series of broad open-ended questions designed to encourage them to talk openly and as spontaneously as possible about their experience of having nasal polyps. In addition, participants were asked more focused questions designed to probe on issues that they may not have mentioned during the course of the interview spontaneously or concepts/statements that required additional clarification. The interviews were transcribed/translated verbatim and qualitative analysis was conducted using Atlas Ti. The symptoms which were most frequently reported spontaneously and were also reported to either be the most frequent, bothersome or worst were categorized as primary symptoms. Number of participants who reported each of the primary symptom is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population included all participants with severe, recurrent nasal polyps enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Nasal congestion | 27
  Breathing difficulties | 27
  Post-nasal drip | 25
  Runny nose | 24
  Head/facial pressure | 23
  Loss of smell | 23
  Ear congestion | 23
  Headache | 23
  Loss of taste | 22

2. Primary Outcome: Number of Participants Who Reported Secondary Symptoms
Description: During the CE section of the interview, participants were asked a series of broad open-ended questions designed to encourage them to talk openly and as spontaneously as possible about their experience of having nasal polyps. In addition, participants were asked more focused questions designed to probe on issues that they may not have mentioned during the course of the interview spontaneously or concepts/statements that required additional clarification. The interviews were transcribed/translated verbatim and qualitative analysis was conducted using Atlas Ti. The symptoms that were reported by fewer participants and less frequently mentioned spontaneously by participants during the interviews were classified as secondary symptoms. Number of participants who reported each of the secondary symptoms is reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Mucus catarrh | 20
  Nose bleeds | 20
  Nasal swelling | 19
  Sneezing | 18
  Nasal pressure | 16
  Nasal pain | 15
  Nasal tightness | 13
  Visible polyps | 6
  Nasal dryness | 7
  Sinus blockage | 18
  Sinus inflammation | 17
  Sinus infections | 16
  Wheezing | 14
  Cough | 19
  Distorted voice | 17
  Dizziness | 16
  Facial pain | 13
  Facial swelling | 9
  Watering eyes | 4
  Visual disturbances | 1
  Itchy eyes | 2
  Red eyes | 1
  Itching ears | 1
  General illness/infection | 4
  Fever | 1

3. Primary Outcome: Number of Participants Who Reported Worst, Most-frequent and Most-bothersome Symptoms
Description: Following spontaneous and probed discussions regarding symptoms during CE interviews, participants were asked to comment on what they each considered to be their 'worst' symptom, their 'most frequent' symptom and their 'most bothersome' symptom. The interviews were transcribed/translated verbatim and qualitative analysis was conducted using Atlas Ti. The number of participants with worst, most-frequent and most-bothersome symptoms are presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Nasal congestion: Worst, n=26: number analyzed (Participants) | 26
  Nasal congestion: Worst, n=26 | 8
  Nasal congestion: most-frequent; n=27 | 9
  Nasal congestion: most bothersome; n=26: number analyzed (Participants) | 26
  Nasal congestion: most bothersome; n=26 | 3
  Difficulty breathing: Worst, n=26: number analyzed (Participants) | 26
  Difficulty breathing: Worst, n=26 | 7
  Difficulty breathing: most-frequent, n=27 | 3
  Difficulty breathing: most bothersome, n=26: number analyzed (Participants) | 26
  Difficulty breathing: most bothersome, n=26 | 7
  Head/facial pressure: Worst, n=26: number analyzed (Participants) | 26
  Head/facial pressure: Worst, n=26 | 6
  Head/facial pressure: most-frequent, n=27 | 6
  Head/facial pressure: most bothersome, n=26: number analyzed (Participants) | 26
  Head/facial pressure: most bothersome, n=26 | 4
  Loss of smell/taste: Worst, n=26: number analyzed (Participants) | 26
  Loss of smell/taste: Worst, n=26 | 3
  Loss of smell/taste: most frequent, n=27 | 1
  Loss of smell/taste: most bothersome, n=26: number analyzed (Participants) | 26
  Loss of smell/taste: most bothersome, n=26 | 2
  Cough: Worst, n=26: number analyzed (Participants) | 26
  Cough: Worst, n=26 | 1
  Cough: most-frequent, n=27 | 1
  Cough: most-bothersome, n=26: number analyzed (Participants) | 26
  Cough: most-bothersome, n=26 | 1
  Nasal discharge: Worst, n=26: number analyzed (Participants) | 26
  Nasal discharge: Worst, n=26 | 1
  Nasal discharge: most-frequent, n=27 | 2
  Nasal discharge: most-bothersome, n=26: number analyzed (Participants) | 26
  Nasal discharge: most-bothersome, n=26 | 0
  Post-nasal drip: Worst, n=26: number analyzed (Participants) | 26
  Post-nasal drip: Worst, n=26 | 1
  Post-nasal drip: most-frequent, n=27 | 2
  Post-nasal drip: most-bothersome, n=26: number analyzed (Participants) | 26
  Post-nasal drip: most-bothersome, n=26 | 5
  Dry mouth: Worst, n=26: number analyzed (Participants) | 26
  Dry mouth: Worst, n=26 | 1
  Dry mouth: most-frequent, n=27 | 0
  Dry mouth: most-bothersome, n=26: number analyzed (Participants) | 26
  Dry mouth: most-bothersome, n=26 | 1
  Painful eyes: Worst, n=26: number analyzed (Participants) | 26
  Painful eyes: Worst, n=26 | 1
  Painful eyes: most-frequent, n=27 | 0
  Painful eyes: most-bothersome, n=26: number analyzed (Participants) | 26
  Painful eyes: most-bothersome, n=26 | 0
  Earache: Worst, n=26: number analyzed (Participants) | 26
  Earache: Worst, n=26 | 1
  Earache: most-frequent, n=27 | 0
  Earache: most-bothersome, n=26: number analyzed (Participants) | 26
  Earache: most-bothersome, n=26 | 0
  Runny nose: Worst, n=26: number analyzed (Participants) | 26
  Runny nose: Worst, n=26 | 0
  Runny nose: most-frequent, n=27 | 1
  Runny nose: most-bothersome, n=26: number analyzed (Participants) | 26
  Runny nose: most-bothersome, n=26 | 3
  Sinus blockage: Worst, n=26: number analyzed (Participants) | 26
  Sinus blockage: Worst, n=26 | 0
  Sinus blockage: most-frequent, n=27 | 1
  Sinus blockage: most-bothersome, n=26: number analyzed (Participants) | 26
  Sinus blockage: most-bothersome, n=26 | 1
  Sneezing: Worst, n=26: number analyzed (Participants) | 26
  Sneezing: Worst, n=26 | 0
  Sneezing: most-frequent, n=27 | 1
  Sneezing: most-bothersome, n=26: number analyzed (Participants) | 26
  Sneezing: most-bothersome, n=26 | 0
  Sinus inflammation: Worst, n=26: number analyzed (Participants) | 26
  Sinus inflammation: Worst, n=26 | 0
  Sinus inflammation: most-frequent, n=27 | 0
  Sinus inflammation: most-bothersome, n=26: number analyzed (Participants) | 26
  Sinus inflammation: most-bothersome, n=26 | 1

4. Primary Outcome: Number of Participants Reporting Proximal Impacts-Physical Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Proximal impacts were defined as those reported to be the direct impact of the symptoms of nasal polyps and included; physical impacts, sleep impacts and impacts on activities of daily living (ADL). The number of participants with physical impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Tiredness/fatigue | 21
  Blowing nose | 19
  Mouth breathing | 14
  Sports/exercise | 14
  Discomfort | 7
  Altered physical appearance | 6
  Mobility | 4
  Increased thirst | 4
  Reduced appetite/weight loss | 2
  Hearing loss | 2
  Spitting mucus | 1
  Smack lips | 1
  Passing out | 1

5. Primary Outcome: Number of Participants Reporting Proximal Impacts-Sleep Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Proximal impacts were defined as those reported to be the direct impact of the symptoms of nasal polyps and included; physical impacts, sleep impacts and impacts on ADL. The number of participants with sleep impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Night-time awakenings | 22
  Poor sleep quality | 12
  Snoring | 11
  Difficulty falling asleep | 9
  Waking partner | 2
  Bedsheet choice | 1
  Comfortable sleep position | 1

6. Primary Outcome: Number of Participants Reporting Proximal Impacts-ADL Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Proximal impacts were defined as those reported to be the direct impact of the symptoms of nasal polyps and included; physical impacts, sleep impacts and impacts on ADL. The number of participants with ADL impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  ADLs affected | 17
  Always being prepared | 8
  Hygiene | 4

7. Primary Outcome: Number of Participants Reporting Distal Impacts-emotional Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Distal impacts were those reported to be impacts of the condition as a whole and included; emotional, social, work/school and treatment impacts. The number of participants with emotional impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Annoyance/frustration | 18
  Sadness | 9
  Irritable/crabby | 9
  Acceptance of nasal polyps | 9
  Stressed | 7
  Scared/worried | 6
  Embarrased | 6
  Loss of enjoyment | 5
  Not understanding condition | 2
  Wanting to be normal | 2
  Isolated | 1
  Worthless | 1
  Not in control | 1
  Suffering | 1
  Not feeling themselves | 1

8. Primary Outcome: Number of Participants Reporting Distal Impacts-social Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Distal impacts were those reported to be impacts of the condition as a whole and included; emotional, social, work/school and treatment impacts. The number of participants with social impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Social activities affected | 12
  Cancelling/avoiding social activities | 12
  Stigma | 7
  Lack of understanding from others | 4
  Improve relationships with family | 3
  Personal relationships affected | 3
  Struggles to hold conversation | 2

9. Primary Outcome: Number of Participants Reporting Distal Impacts-work/School Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Distal impacts were those reported to be impacts of the condition as a whole and included; emotional, social, work/school and treatment impacts. The number of participants with work/school impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Time off work | 17
  Affects activities at work | 10
  Reduced productivity | 5
  Inability to focus | 5
  Taking breaks | 4
  Symptom triggers in the workplace | 3
  Loss of income | 3
  Fatigue at work | 3
  Reduced smell at work | 3
  Blowing nose at work | 3

10. Primary Outcome: Number of Participants Reporting Distal Impacts-treatment Impact
Description: The impacts as reported by participants during CE interviews were categorized as proximal impacts and distal impacts. Distal impacts were those reported to be impacts of the condition as a whole and included; emotional, social, work/school and treatment impacts. The number of participants with treatment impacts are reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Cost of treatment | 7
  Short treatment efficacy | 7
  Side effects of medication | 5
  Lack of treatment efficacy | 2
  Fear of taking medication | 2

11. Primary Outcome: Number of Participants Who Reported Symptoms to be Targeted by New Treatment
Description: During CE interviews, participants were asked about the changes they would like to see from a new treatment for nasal polyps and which symptoms would be most meaningful for the treatment to target. The number of participants with their reported symptoms to be targeted by new treatment is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who were asked about treatment preferences were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 24
Participants
  Nasal congestion | 12
  Breathing difficulty | 8
  Head/facial pressure | 5
  Post-nasal drip | 4
  Loss of taste | 4
  Loss of smell | 2
  Headache | 2
  Ear pressure | 1
  Dizziness | 1

12. Primary Outcome: Number of Participant Who Reported Impacts to be Targeted by New Treatment
Description: During CE interviews, participants were asked about the changes they would like to see from a new treatment for nasal polyps and which impacts would be most meaningful for the treatment to target. The number of participants with corresponding impacts to be targeted by new treatment is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who were asked about treatment preferences were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 24
Participants
  Reduction in need for surgery & in polyp regrowth | 6
  Ability to do physical activity | 3
  Sleep disturbance | 3
  Less need for medications | 2
  Regain energy | 1
  Able to concentrate | 1
  Dry mouth | 1
  Able to blow nose | 1

13. Primary Outcome: Number of Participants Reporting Factors to be Considered for Surgery
Description: During CE interviews, participants were asked about experiences of their surgery in past. The number of participants with the corresponding factors to be considered for surgery is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who discussed the factors were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 26
Participants
  Seriousness of surgery | 3
  Success of surgery | 3
  Unable to bear symptoms any longer | 3
  Confidence in doctor | 3
  Treatment failure | 3
  Simplicity of surgery | 3
  No alternative | 2
  Own research | 1
  Age | 1
  Pain/recovery | 1
  Risk of surgery | 1
  Risk of scarring | 1
  Life expectancy | 1

14. Primary Outcome: Number of Participants With Ease of Decision to Have Surgery
Description: During CE interviews, participants were asked about experiences of their surgery in past. The number of participants with ease of decision to have surgery is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Decision was easy | 6
  Decision was difficult | 6

15. Primary Outcome: Number of Participants Who Reported on the Positive or Negative Impacts of Surgery
Description: During CE interviews, participants were asked about experiences of their surgery in past. The number of participants who reported on the positive or negative impacts of surgery is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Positive impact of surgery | 21
  Negative impact of surgery | 23

16. Primary Outcome: Number of Participants Who Did Not Understand Visual Analog Scale (VAS) Assessment
Description: Participants were required to complete six VAS assessments (overall symptom VAS and single item VAS) as a part of the CD interview. The participants evaluated their overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 centimeter (cm) or 100 millimeter (mm) whereby 0 represents 'no symptom' and 10 or 100 represents 'as bad as you can imagine' respectively. Participants were asked to speak aloud their thoughts as they read the instructions and completed the questions. After completion of each think-aloud exercise, participants were also probed upon their understanding of the instrument items. Number of participants who did not understand the VAS assessments is reported.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Overall symptoms | 0
  Facial pain/pressure | 0
  Loss of smell | 0
  Mucus in the throat | 0
  Nasal discharge | 1
  Nasal obstruction | 0

17. Primary Outcome: Number of Participants Who Reported Symptoms Assessed by VAS to be Relevant to Their Condition
Description: Participants were required to complete six VAS assessments (overall symptom VAS and single item VAS) as a part of the CD interview. The participants evaluated their overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 cm or 100 mm whereby 0 represents 'no symptom' and 10 or 100 represents 'as bad as you can imagine' respectively. Participants were asked to speak aloud their thoughts as they read the instructions and completed the questions. After completion of each think-aloud exercise, participants were also probed about the relevance of VAS items. Relevance was determined based on participants personal descriptions and related discussion of their experience of each symptom or impact during CD interview. It was also determined via the rating of a given symptom/impact on each measure as greater than a score of zero. Number of participants who reported the symptoms assessed by VAS to be relevant are presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Overall symptoms | 26
  Facial pain/pressure | 25
  Loss of smell | 24
  Mucus in the throat | 25
  Nasal discharge | 26
  Nasal obstruction | 25

18. Primary Outcome: Number of Participants Who Liked or Disliked VAS Assessments
Description: Participants were required to complete six VAS assessments (overall symptom VAS and single item VAS) as a part of the CD interview. The participants evaluated their overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 cm or 100 mm whereby 0 represents 'no symptom' and 10 or 100 represents 'as bad as you can imagine' respectively. Participants provided a general feedback on completing the six VAS assessments which included relevance of symptoms to their condition, ease of completion and interpretation of the scale. The number of participants who provided general feedback for VAS assessments in terms of likes or dislikes for VAS assessment is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who provided general feedback were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 26
Participants
  VAS likes | 17
  VAS dislikes | 2

19. Primary Outcome: Number of Participants With Difficulties Completing VAS Assessments
Description: Participants were required to complete six VAS assessments (overall symptom VAS and single item VAS) as a part of the CD interview. The participants evaluated their overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 cm or 100 mm whereby 0 represents 'no symptom' and 10 or 100 represents 'as bad as you can imagine' respectively. Participants provided a general feedback on completing the six VAS assessments which included relevance of symptoms to their condition, ease of completion and interpretation of the scale. The number of participants with difficulties completing VAS assessment is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who provided general feedback were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 26
Participants | 7

20. Primary Outcome: Number of Participants Who Understood VAS Anchors
Description: Participants completed the VAS assessment as a part of the CD interview. Participants evaluated their overall symptom severity, or the severity of individual symptoms of nasal polyps along a continuum, typically of 10 cm or 100 mm whereby 0 represents 'no symptom' and 10 or 100 represents 'as bad as you can imagine' respectively. Participants were asked about their understanding of the response continuum for VAS assessment. Number of participants who understood the VAS anchors (100 as bad as you can imagine and 0 none) is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants with data available at the specified time points were included in the analysis (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  100=as bad as you can imagine; n=27 | 27
  0=none; n=24: number analyzed (Participants) | 24
  0=none; n=24 | 23

21. Primary Outcome: Number of Participants Who Did Not Understand the Items of Sino-nasal Outcomes Test (SNOT)-22
Description: Participants completed SNOT-22 assessment as a part of the CD interview. The SNOT-22 contains 22 nose, sinus, and general health-related quality of life (HRQoL) items and is used to measure HRQoL associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Number of participants who did not understand the items of SNOT-22 is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who were asked about each item was analyzed (represented by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Need to blow nose; n=25: number analyzed (Participants) | 25
  Need to blow nose; n=25 | 0
  Nasal blockage; n=27 | 0
  Sneezing; n=26: number analyzed (Participants) | 26
  Sneezing; n=26 | 1
  Runny nose; n=25: number analyzed (Participants) | 25
  Runny nose; n=25 | 3
  Cough; n=26: number analyzed (Participants) | 26
  Cough; n=26 | 0
  Post-nasal discharge; n=27 | 4
  Thick nasal discharge; n=26: number analyzed (Participants) | 26
  Thick nasal discharge; n=26 | 2
  Ear fullness; n=27 | 1
  Dizziness; n=27 | 0
  Ear pain; n=23: number analyzed (Participants) | 23
  Ear pain; n=23 | 0
  Facial pain/pressure; n=25: number analyzed (Participants) | 25
  Facial pain/pressure; n=25 | 0
  Decreased sense of smell/taste; n=27 | 0
  Difficulty falling asleep; n=27 | 0
  Wake up at night; n=27 | 0
  Lack of good night's sleep; n=24: number analyzed (Participants) | 24
  Lack of good night's sleep; n=24 | 1
  Wake up tired; n=25: number analyzed (Participants) | 25
  Wake up tired; n=25 | 0
  Fatigue; n=24: number analyzed (Participants) | 24
  Fatigue; n=24 | 0
  Reduced productivity; n=26: number analyzed (Participants) | 26
  Reduced productivity; n=26 | 0
  Reduced concentration; n=26: number analyzed (Participants) | 26
  Reduced concentration; n=26 | 0
  Frustration/restless/irritable; n=26: number analyzed (Participants) | 26
  Frustration/restless/irritable; n=26 | 0
  Sad; n=26: number analyzed (Participants) | 26
  Sad; n=26 | 1
  Embarrassed; n=26: number analyzed (Participants) | 26
  Embarrassed; n=26 | 1

22. Primary Outcome: Number of Participants Who Reported Symptoms Assessed by SNOT-22 as Relevant to Their Condition
Description: Participants were required to complete SNOT-22 assessment as a part of the CD interview. The SNOT-22 contains 22 nose, sinus, and general HRQoL items and is used to measure health-related quality of life associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Number of participants who reported the symptoms assessed by SNOT-22 to be relevant to their condition are presented.
Time Frame: Up to 120 minutes
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants
  Need to blow nose; n=27 | 25
  Nasal blockage; n=25: number analyzed (Participants) | 25
  Nasal blockage; n=25 | 24
  Sneezing; n=25: number analyzed (Participants) | 25
  Sneezing; n=25 | 20
  Runny nose; n=26: number analyzed (Participants) | 26
  Runny nose; n=26 | 22
  Cough; n=25: number analyzed (Participants) | 25
  Cough; n=25 | 19
  Post-nasal discharge; n=23: number analyzed (Participants) | 23
  Post-nasal discharge; n=23 | 20
  Thick nasal discharge; n=23: number analyzed (Participants) | 23
  Thick nasal discharge; n=23 | 20
  Ear fullness; n=27 | 21
  Dizziness; n=25: number analyzed (Participants) | 25
  Dizziness; n=25 | 15
  Ear pain; n=26: number analyzed (Participants) | 26
  Ear pain; n=26 | 16
  Facial pain/pressure; n=24: number analyzed (Participants) | 24
  Facial pain/pressure; n=24 | 22
  Decreased sense of smell/taste; n=23: number analyzed (Participants) | 23
  Decreased sense of smell/taste; n=23 | 18
  Difficulty falling asleep; n=26: number analyzed (Participants) | 26
  Difficulty falling asleep; n=26 | 21
  Wake up at night; n=27 | 25
  Lack of good night's sleep; n=22: number analyzed (Participants) | 22
  Lack of good night's sleep; n=22 | 19
  Wake up tired; n=25: number analyzed (Participants) | 25
  Wake up tired; n=25 | 21
  Fatigue; n=27 | 22
  Reduced productivity; n=26: number analyzed (Participants) | 26
  Reduced productivity; n=26 | 21
  Reduced concentration; n=25: number analyzed (Participants) | 25
  Reduced concentration; n=25 | 21
  Frustration/restless/irritable; n=23: number analyzed (Participants) | 23
  Frustration/restless/irritable; n=23 | 19
  Sad; n=26: number analyzed (Participants) | 26
  Sad; n=26 | 15
  Embarrassed; n=26: number analyzed (Participants) | 26
  Embarrassed; n=26 | 16

23. Primary Outcome: Number of Participants Who Liked or Disliked SNOT-22 Assessments
Description: The SNOT-22 contains 22 nose, sinus, and general HRQoL items and is used to measure health-related quality of life associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Participants provided a general feedback on completing the SNOT-22 which included relevance of symptoms to their condition, ease of completion and interpretation of the scale. Number of participants who liked or disliked the SNOT-22 is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who provided general feedback were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 24
Participants
  SNOT-22 likes | 11
  SNOT-22 dislikes | 9

24. Primary Outcome: Number of Participants With Difficulties Completing SNOT-22
Description: Participants provided a general feedback on completing the SNOT-22 during the CD interview. The SNOT-22 contains 22 nose, sinus, and general HRQoL items and is used to measure health-related quality of life associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Number of participants with difficulties completing SNOT-22 assessment is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who were interviewed for ease of completion were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 20
Participants | 3

25. Primary Outcome: Number of Participants Who Understood SNOT-22 Response Options
Description: Participants completed SNOT-22 as a part of the CD interview. The SNOT-22 contains 22 nose, sinus, and general HRQoL items and is used to measure health-related quality of life associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Participants were asked about their understanding of each of the six options (no problem, mild or slight problem, very mild problem, moderate problem, severe problem, as bad as it can be) included in SNOT-22. Number of participants who understood each of the six SNOT-22 response options is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 27
Participants | 27

26. Primary Outcome: Number of Participants Who Reported Missing SNOT-22 Items
Description: Participants completed SNOT-22 as a part of the CD interview. The SNOT-22 contains 22 nose, sinus, and general HRQoL items and is used to measure health-related quality of life associated with rhinosinusitis with or without nasal polyps. Within the SNOT-22, participants were required to indicate the level to which each listed nasal, sinus or HRQoL experience has been affected on a 6-point scale ranging from 0 (No problem) to 5 (Problem as bad as it can be). Participants were asked if they felt any items were missing from SNOT-22. Number of participants who reported missing items in SNOT-22 is presented.
Time Frame: Up to 120 minutes
Population: All Enrolled Population. Only those participants who were asked about missing items were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 14
Participants | 5

27. Secondary Outcome: Number of Participants Reporting Symptom Variability-Application (App) Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Participants completed a number of tasks across 10 days, which explored how nasal polyp symptoms and impacts varied across a full day (within day variability) or assess the day to day variability (between day variability). Number of participants reporting within day and between-day symptom variability is reported.
Time Frame: Up to 10 days
Population: All Enrolled Population. Only those participants who took part in the real-world data capture activity were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Within day variability | 9
  Between-day variability | 7

28. Secondary Outcome: Number of Participants Reporting Primary Symptoms as Identified During App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting primary symptoms as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Nasal congestion | 8
  Difficulty breathing | 8
  Head/facial pressure | 7
  Post-nasal drip | 6
  Runny nose | 6
  Loss of smell | 5
  Loss of taste | 4

29. Secondary Outcome: Number of Participants Reporting Secondary Symptoms as Identified During App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting secondary symptoms as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Nasal swelling | 3
  Nasal pain | 3
  Sneezing | 2
  Nasal dryness | 2
  Nasal tightness | 1
  Nasal itching | 1
  Nasal burning | 1
  Nasal scabs | 1
  Sinus inflammation | 1
  Sinus infection | 1
  Throat pain | 1
  Cough | 2
  Distorted voice | 3
  Face swelling | 5
  Facial pain | 3
  Dizziness | 3
  Headache | 4
  Ear pain | 1
  Watering eyes | 1
  Nasal tingling | 1
  Illness/infection | 1

30. Secondary Outcome: Number of Participants Reporting Physical Impacts as Idenfied During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants with physical impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Blowing nose | 5
  Breathing through mouth | 5
  Dry throat/mouth | 5
  Tiredness/fatigue | 3
  Thirst | 3
  Discomfort | 3
  Physical activity difficulties | 2
  Altered physical appearance | 1
  Hearing loss | 1

31. Secondary Outcome: Number of Participants Reporting Sleep Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting sleep impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Waking up at night | 3
  Difficulty finding comfortable sleep position | 3
  Difficulty falling asleep | 2
  General poor sleep quality | 2
  Snoring | 1

32. Secondary Outcome: Number of Participants Reporting ADL Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting ADL impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Restricts activities of daily living | 3
  Unpredictably of condition | 1
  Hygiene | 1

33. Secondary Outcome: Number of Participants Reporting Emotional Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting emotional impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Embarrassment | 4
  Sadness | 3
  Anger | 3
  Irritable | 3
  Stressed | 1

34. Secondary Outcome: Number of Participants Reporting Social Functioning Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting social functioning impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Social isolation | 1
  Impacts personal relationships | 1

35. Secondary Outcome: Number of Participants Reporting Work Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting work impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Certain work activities affected | 2
  Reduced productivity | 1
  Reduced concentration | 1

36. Secondary Outcome: Number of Participants Reporting Treatment Impacts as Identified During the App Task
Description: Participants took part in an app-based real-world data capture activity. The participants were required to download an app to their smart phone or tablet. Data capture was conducted over a 10-day period during which participants were required to complete a series of questions/tasks via the smartphone/tablet application in real-time. The questions/tasks were designed to explore the experience of nasal polyps. Participants provided responses to the questions using a variety of methodologies including video, audio, text and photographic responses with captions. Number of participants reporting treatment impacts as identified during app task is reported.
Time Frame: Up to 10 days
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Interview Participants With Nasal Polyps
Number analyzed (Participants) | 10
Participants
  Side effects of medications | 3
  Lack of efficacy | 2
  Short efficacy | 2
  Overwhelming number of medications | 2
  Cost of medications | 1

ADVERSE EVENTS:
Time Frame: Up to 10 days
Description: AEs and SAEs were observed in All Enrolled Population.
Arm/Group | Interview Participants With Nasal Polyps
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT03221192/Prot_SAP_ICF_000.pdf